CLINICAL TRIAL: NCT03811223
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Crossover Trial to Evaluate the Effects of Evolocumab Added to Standard Lipid-lowering Therapy on Fasting and Post Fat Load Lipids in Patients With Familial Dysbetalipoproteinemia
Brief Title: Effects of Evolocumab Versus Placebo Added to Standard Lipid-lowering Therapy on Fasting and Post Fat Load Lipids in Patients With Familial Dysbetalipoproteinemia
Acronym: EVOLVE-FD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, dr.Frank L.J. Visseren, prof. dr. F.L.J. Visseren, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCU-VASC-CO-002
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Familial Dysbetalipoproteinemia; Hyperlipoproteinemia Type III
Keywords: Postprandial hyperlipidemia; Evolocumab; PCSK9 monoclonal antibody
MeSH Terms: conditions — Hyperlipoproteinemia Type III | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Experimental): Evolocumab 140 mg subcutaneous injection once every 2 weeks for 12 weeks
  Interventions: Drug: Evolocumab Auto-Injector [Repatha]
- Placebo (Placebo Comparator): Placebo injection once every 2 weeks for 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Evolocumab Auto-Injector [Repatha] — Evolocumab 140 mg every 2 weeks for 12 weeks
  Arms: Evolocumab
Drug: Placebos — Placebo subcutaneous injection every 2 weeks for 12 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Patients with familial dysbetalipoproteinemia (FD) have increased triglycerides, non-high-density lipoprotein cholesterol (non-HDL-C), beta VLDL, premature atherosclerosis and cardiovascular disease. They also have a delayed postprandial triglyceride and chylomicron (CM) remnant clearance. Postprandial hypertriglyceridemia is associated with increased vascular risk. Although combination therapy with statin and fibrate is recommended in the treatment of patients with FD, there is still a substantial amount of patient who do not reach their treatment target with this medication. Furthermore no information is available about the postprandial effects of adding evocolumab to standard lipid lowering therapy in FD patients.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed with Familial Dysbetalipoproteinemia;

   * ε2ε2 genotype or dominant APOE mutation genotype (confirmed by genotyping or isoelectric focusing) with any lipid-lowering treatment at a stable dose for at least three months and non-HDL-C >1.6 mmol/L or;
   * Patients with ε2ε2 genotype or dominant APOE mutation (confirmed by genotyping or isoelectric focusing) without lipid-lowering treatment and with an ApoB/TC ratio < 0.15.
2. >18 years old (on the day of signing informed consent).
3. Women are postmenopausal and not receiving hormone therapy (including cyclic and non-cyclical hormone replacement therapy or any estrogen antagonist/agonist). Postmenopausal status is defined as:

   * no menses for ≥3 years or;
   * no menses for ≥1 year but <3 years and confirmed by FSH levels elevated into the postmenopausal range (15-150 IU/L).
4. Willingness to maintain a stable diet for the duration of the study.
5. Understanding of the study procedures, alternative treatments available, and risks involved with the study and voluntarily agreement to participate by giving written informed consent.

Exclusion criteria:

1. Intolerance, known allergy or hypersensitivity to evolocumab (or other PCSK-9 monoclonal antibodies), latex or any of the components of the medication.
2. Current or prior exposure to evolocumab or another PCSK9-inhibitor mAb in the past 12 weeks.
3. Unable or unwilling to drink an oral fat load.
4. Premenopausal women.
5. Uncontrolled diabetes as defined by a HbA1c >69 mmol/mol.
6. BMI >40 kg/m2.
7. Uncontrolled blood pressure with systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg.
8. Increased hepatic enzymes, defined as alanine transaminase (ALAT) or aspartate transaminase (ASAT) >3 times the ULN, or active liver disease defined as non alcoholic steatohepatitis (NASH), cirrhosis or Child Pugh B and C, or history of chronic active hepatitis B or C; subjects with documented resolution after treatment are permitted.
9. Impaired renal function, defined by an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2, and/or need of renal placement therapy or other clinically significant renal disease.
10. (Sub)clinical hypothyroidism defined as TSH >5.0 mcl/U/mL or (sub)clinical hyperthyroidism defined as TSH < 0.35 mcl/U/ml.
11. Increased levels of creatinine kinase defined as >3 times the ULN.
12. Increased fasting levels of triglycerides defined as >10 mmol/L.
13. History of organ transplantation and/or use of immunosuppressive medication.
14. Use of fish oil or red yeast rice, bempedoic acid, niacin, CETP inhibitors, lomitapide, mipomersen < 6 weeks prior to the study or the use of siRNA targeting PCSK9 inhibitors < 36 weeks prior to the study.
15. Active malignancy (<2 year prior to informed consent), except non-melanoma skin cancer or carcinoma in situ of the cervix.
16. Known infection with Human Immunodeficiency Virus (HIV) or AIDS.
17. Known celiac disease or other disorder associated with significant intestinal malabsorption.
18. Known galactose-intolerance, Lapp-lactase deficiency or glucose-galactose malabsorption.
19. Alcohol use, defined as >14 alcoholic consumptions per week for women and >21 alcohol consumptions per week for men. One alcohol consumption unit is defined as follows: 350 mL beer, 150 mL wine or 45 mL alcohol for mixed drinks.
20. Current participation or participation in a study with an investigational compound or device within 30 days of signing informed consent.
21. Any medical, social or physiological circumstance which interferes the study, based on judgement by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
AUC (area under the curve) non-HDL-cholesterol | 12 weeks

SECONDARY OUTCOMES:
Fasting levels, AUC and iAUC of total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides and ApoB, as well as fasting non-HDL-cholesterol. | 12 weeks
Percentage change from baseline and absolute difference in fasting and post fat load non-HDL-cholesterol, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides and ApoB. | 12 weeks
Fasting and post fat load lipoprotein (VLDL1, VLDL2, IDL, LDL, HDL) concentrations and composition (triglycerides, cholesterol, ApoB and apolipoproteins). | 12 weeks
Post fat load ApoB 48-containing lipoprotein concentrations (chylomicrons and chylomicron remnants) and proteins involved in postprandial lipid metabolism. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank LJ Visseren, prof, Principal Investigator — UMC Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there is no plan to make individual participant data available to other researchers, but this is possible in the future.